CLINICAL TRIAL: NCT04086966
Title: PSMA-PET/MRI for Radiation Treatment Planning in Patients With Locally Metastatic Prostate Cancer: A Pilot Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Samuel Joseph Galgano, Program Director, Abdominal Imaging Fellowship Assistant Professor, Abdominal Imaging Section and Division of Molecular Imaging and Therapeutics, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R18-190 IRB-300003826
Record Dates: First submitted 2019-09-09; First posted 2019-09-12 (Actual); Results first posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2023-11

CONDITIONS: Metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Metastatic Prostate Cancer Arm (Experimental): [68Ga]PSMA-11 PET/MRI or PET/CT for guiding the radiation treatment plan in patients with known or suspected locally metastatic prostate cancer
  Interventions: Drug: [68Ga]PSMA-PET/MRI or PET/CT

INTERVENTIONS:
Drug: [68Ga]PSMA-PET/MRI or PET/CT — [68Ga]PSMA-PET/MRI or PET/CT

SUMMARY:
This pilot study will investigate the use of PSMA-PET/MRI (Positron Emission Tomography/ Magnetic Resonance Imaging)to guide radiation treatment planning in patients with known or suspected locally metastatic prostate cancer at the time of diagnosis. Patients will undergo a single PSMA-PET/MRI (or PET/CT (Computed Tomography) in some circumstances) prior to initiation of treatment. Following development of a PSMA-PET guided radiation treatment plan, therapeutic radiation will be delivered per standard-of-care parameters and assessments of feasibility and tolerability will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven treatment-naïve prostate adenocarcinoma with pelvic metastases known to suspected on standard-of-care staging imaging
* Eligibility and plan to undergo definitive radiation therapy for prostate cancer per established standard-of-care radiation oncology clinical guidelines
* Be at least 18 years of age

Exclusion Criteria:

* Inability to tolerate or undergo PET/MRI or PET/CT
* Previous or current hematologic or lymphatic disorder (including leukemia, lymphoma, Castleman's disease, etc.)
* Recurrent prostate adenocarcinoma
* Known distant metastatic disease
* Current or prior treatment for prostate cancer
* Known allergy to glucagon
* Previous diagnosis of insulinoma or pheochromocytoma

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2022-02-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham Medical Center, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Metastatic Prostate Cancer Arm
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Metastatic Prostate Cancer Arm
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients Who Demonstrate Pelvic Lymph Node Metastases on PSMA-PET/MRI That Were Not Detected on MRI
Time Frame: 1 scan
Measure: Count of Participants; unit: Participants
Arm/Group | Metastatic Prostate Cancer Arm
Number analyzed (Participants) | 10
Participants | 3

2. Secondary Outcome: The Total Number of Pelvic Nodal Metastases Detected on PSMA-PET/MRI
Time Frame: 1 scan
Measure: Number; unit: lymph nodes
Arm/Group | Metastatic Prostate Cancer Arm
Number analyzed (Participants) | 10
lymph nodes | 19

3. Secondary Outcome: Number of Patients in Whom Dose-escalated Radiotherapy Can be Feasibly Delivered
Time Frame: 1 simulation scan
Measure: Count of Participants; unit: Participants
Arm/Group | Metastatic Prostate Cancer Arm
Number analyzed (Participants) | 10
Participants | 8

4. Secondary Outcome: Number of Patients Who Experience CTCAE (Common Terminology Criteria for Adverse Events) Grade 3-5 GI or GU Toxicities
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Metastatic Prostate Cancer Arm
Number analyzed (Participants) | 10
Participants | 0

5. Secondary Outcome: The Total Number of Pelvic Nodal Metastases Detected on MRI
Time Frame: 1 scan
Measure: Number; unit: lymph nodes
Arm/Group | Metastatic Prostate Cancer Arm
Number analyzed (Participants) | 10
lymph nodes | 9

ADVERSE EVENTS:
Time Frame: 18 months
Description: Standard CTCAE assessment during radiation therapy
Arm/Group | Metastatic Prostate Cancer Arm
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-15): https://cdn.clinicaltrials.gov/large-docs/66/NCT04086966/Prot_SAP_000.pdf